CLINICAL TRIAL: NCT00585273
Title: Cardiovascular Complications of First-line, Second-generation Antipsychotics
Brief Title: Antipsychotics and Blood Vessel Function
Status: Completed | Type: Observational
Sponsor: Jess G. Fiedorowicz (Other)
Responsible Party: Sponsor-Investigator, Jess G. Fiedorowicz, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 200703764; University of Iowa GCRC #0740
Record Dates: First submitted 2007-12-19; First posted 2008-01-03 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Bipolar Disorder; Schizophrenia
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Incident users of antipsychotics.
- 2: Non-users of antipsychotics

SUMMARY:
Over the last decade, second generation antipsychotics have been increasingly utilized. Since their introduction, however, atypical antipsychotics have been increasingly associated with significant metabolic complications including hyperlipidemia, insulin resistance/diabetes mellitus, and obesity. These metabolic complications increase the risk for cardiovascular disease in populations with an already elevated risk.

The initial goal of the proposed study is to identify early signs of endothelial dysfunction and vascular disease in those treated with atypical antipsychotics. The identification of early signs of vascular disease may further link metabolic complications with any cardiovascular risk. Demonstration of changes in vascular function associated with atypical antipsychotics represents an important identifiable intermediate of more long-term cardiovascular risk.

The second goal of the proposed study is to identify genetic factors that may be associated with the development of cardiovascular disease, which can later serve as a guide to predict risk. Accurate prediction of risk may facilitate the future development of an empirical, risk-based, individualized selection process for antipsychotic medications.

Aim 1: To quantify the role of antipsychotic-induced metabolic complications on the development of vascular disease using measures of endothelial function.

Hypothesis 1: Atypical antipsychotics will lead to greater impairments in endothelial function, evidenced by decreased flow-mediated dilation from baseline measures and compared with changes over time in controls. Medication-induced metabolic complications will be temporally associated with these impairments in endothelial function.

Aim 2: To investigate the role of candidate pharmacogenetic polymorphisms with cardiovascular and metabolic complications of atypical antipsychotics.

Hypothesis 2: Profiles of polymorphisms at receptors targeted by atypical antipsychotics will be associated with impaired cardiovascular function and metabolic complications.

DETAILED DESCRIPTION:
Participants will have all evaluations related to metabolic complications performed in the University of Iowa Clinical Research Unit (CRU) or in the EndoPAT laboratory located in Room 269 GH. For all visits, weights will be measured without shoes, in light clothing, using an electronic scale that measures to the nearest 0.25 kg. Standing heights will be measured without shoes, to the nearest 0.1 cm using a free-standing stadiometer. These weights and heights will be utilized for the computation of body mass index (BMI). Waist circumference will be measured horizontally at the tip of the right iliac crest in the standing position using a measuring tape. Blood pressure and heart rate will be measured in the sitting position after five minutes of silent rest, using an automated sphygmomanometer. An ambulatory blood pressure will also be obtained at each visit. An EKG will be conducted during Visit 1. Dual energy X-ray absortionmetry (DEXA) will assess percentage of body fat at intake, Visit 4 and Visit 8. If a participant is unable to complete a DEXA scan, body fat will be determined using the BOD POD® Gold Standard Body Composition Tracking System. The BOD POD® is an integrated system consisting of a digital scale to measure subject mass, a large egg-shaped fiberglass air displacement plethysmography (ADP) to determine body volume (BV), and a computer that operates the equipment and calculates body composition. Body density is determined from subject mass and volume measurements and then percent fat is calculated using one of several standard formulas. CRU dieticians will perform skin fold measurements at intake and completion. Fasting measures of triglycerides, LDL-C, HDL-C, IDL, VLDL, apolipoprotein A, apolipoprotein B, Lp(a) cholesterol, C-reactive protein, IL-6, leptin levels, insulin levels, and glucose will be obtained at baseline, 2 weeks, 12 weeks, 26 weeks, 1 year, 2 years, 3 years and 4 years. Hemoglobin A1C will be collected at baseline and weeks 12 and 26, 1 year, 2 years, 3 years and 4 years. Cholesterol levels will be determined by an enzymatic calorimetric test using cholesterol esterase and cholesterol oxidase. LDL-C and HDL-C fractions will be obtained via a homogeneous enzymatic in vitro colorimetric assay. For the determination of triglyceride levels, free glycerol is eliminated prior to hydrolysis of triglycerides in a preliminary reaction where lipase and 4-aminophenazone are omitted, followed by enzymatic hydrolysis of triglycerides and determination of the liberated glycerol by a fully enzymatic colorimetric assay reaction. Apolipoproteins and other lipid parameters will be measured using beta quantification through the Mayo Medical Laboratories (unit code 83673).

Endothelial and Cardiovascular Function: Participants will have endothelial function measured at baseline, and each subsequent visit. To maximize completion rates, participants planning to discontinue their antipsychotic between weeks 16 and 26 will have their final measures taken at the time of discontinuation. Prior to these appointments, participants will be instructed to not eat or drink anything (including caffeinated products such as coffee, tea, soda, etc.) except water for at least 12 hours prior to the appointment. They will also be instructed to not drink any alcohol for 24 hours prior to each study. They will be asked not to smoke for the two hours prior to the study. Administration of blood pressure and lipid lowering medications for that day will be delayed until after the procedures. Measures of endothelial function will be obtained in the Clinical Research Unit (CRU).

CONDUIT VESSEL FUNCTION: Conduit vessel endothelial function will be assessed non-invasively via ultrasound measurement of brachial artery diameter during changes in brachial artery flow. The technique uses a 10-13 MHz linear array transducer ultrasound system (Biosound ESAOTE, Indianapolis, IN). A 5 cm length of the brachial artery is imaged in longitudinal section above the antecubital fossa and the optimal probe site on the skin marked. Baseline images of brachial artery diameter and Doppler velocities from the center of the vessel are recorded on videotape. While images for brachial artery diameter are being continuously recorded, an occluding forearm cuff placed just below the antecubital fossa is inflated for 5 minutes. The brachial artery diameter and Doppler velocities are continuously recorded before, during and after cuff deflation. After approximately 5 minutes, once basal diameter and flow have been restored, nitroglycerin (300 mcg) will be administered sublingually and measurements made for an additional 6 minutes.

HEART RATE AND BLOOD PRESSURE VARIABILITY: We will also assess blood pressure and heart rate variability using recordings of indirect arterial pressure with a beat-to-beat finger systolic and diastolic blood pressure recording in conjunction with the electrocardiogram tracing during the conduit vessel function procedures. Data from this measurement will allow us to assess blood pressure and heart rate variability. Cardiovascular variability (HRV) is a marker for cardiovascular risk whereby lower variability indicates greater risk for myocardial infarct and stroke. This procedure can be performed during assessment of conduit vessel function so requires no additional time.

ARTERIAL TONOMETRY: We will utilize arterial tonometry through measurement of pulse wave analysis (PWA) and pulse wave velocity (PWV) using a SphygmorCor machine. This machine uses a noninvasive probe, pressed lightly on the skin over the carotid, radial and femoral arteries for about five minutes each. These measurements will provide a measure of arterial compliance, stiffness, and other hemodynamic information. The PWA system is a computerized diagnostic tool for the assessment of central blood pressure. The peripheral pressure pulse waveform contains information in addition to the maximum and minimal values (systolic and diastolic pressures). The PWA system can derive the central aortic pressure waveform from the peripheral pressure waveform recorded at the radial or carotid arteries. The system uses mathematical transforms to derive the central aortic pressure pulse waveform and then calculates a range of central indices of ventricular-vascular interaction, which are displayed both graphically and numerically. The PWV system measures the velocity of the blood pressure waveform between any two superficial artery sites. A pressure tonometer is used to transcutaneously record the pressure pulse waveforms in the underlying artery. The pressure pulse waveform is recorded simultaneously with an electrocardiogram (ECG) signal, which provides an R-wave timing reference. Pressure pulse recordings are performed consecutively at the two superficial artery sites over the carotid and femoral artery. The software processes each set of pressure pulse and ECG waveform data to calculate the mean time difference between the R-wave and the pressure wave- on a beat-by-beat basis. The PWV is then calculated using the mean time difference and the arterial path length between the two recording sites. The velocity of the blood pressure pulse waveform is dependent on the stiffness of the artery along which the pulse is traveling. Serial measurement of pulse wave velocity in a section of artery will indicate the magnitude of change in arterial stiffness in that section of the artery.

PSYCHIATRIC ASSESSMENT: Detailed historical information will be gathered including age, occupation, education, race, height, weight, medical history, treatment history, family history of medical illness with focus on risk factors for metabolic syndrome, and substance use history including tobacco. Basic clinical information will be obtained to verify psychiatric diagnosis and assess cardiac risk by the Framingham Heart Study formula. It is estimated that this history will take 45 minutes to complete. Affective and psychotic symptomatology will be cross-sectionally assessed using the Montgomery Asberg Depression Rating Scale, the Young Mania Scale, and the Brief Psychotic Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Being started on a first-line, second-generation, antipsychotic associated with weight gain (risperidone, olanzapine, or quetiapine) for the treatment of an affective or psychotic disorder -OR- psychiatric controls not taking antipsychotic medications will also be enrolled

Exclusion Criteria:

* Exclusion criteria will include the presence of any of the following: neoplasm, active thyroid disease (i.e. not euthyroid), pregnancy or planned pregnancy, diabetes mellitus, Raynaud's disease, anticoagulant therapy, or inability to provide informed consent. We will exclude participants who have started valproic acid derivatives in the preceding 6 months, given its association with insulin resistance and weight gain. Participants with active substance abuse or dependence will also be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Thirty patients, 18 - 50 years of age, who are being started on a first-line, second-generation, antipsychotic associated with weight gain (risperidone, olanzapine, or quetiapine) for the treatment of an affective or psychotic disorder, will be invited to participate. Participants must not have taken any of these antipsychotics or clozapine in the preceding three months. Another twenty psychiatric controls not taking antipsychotic medications will also be enrolled. Statistically, controls will serve primarily to compare changes in flow-mediated dilation over time rather than for direct comparison of variables between groups. Participation will be voluntary and initiated upon clinician or self-referral.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2007-09; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation | 6 months
  % dilation of the brachial artery in response to 5 minutes of ischemia
Forearm vascular resistance | 6 months
  % dilation of forearm blood vessels in response to pharmacological challenge measured using plethysmography

CONTACTS AND LOCATIONS:
Overall Officials: Jess G Fiedorowicz, M.D., Ph.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for de-identified data may be presented to the principal investigator with a statistical analysis plan.
Time Frame: Data will be made available on 8/27/2019 for a period of at least three years.
Access Criteria: Requests for data will be reviewed by Principal Investigator Jess Fiedorowicz for additional analyses provided a statistical analysis plan.

REFERENCES:
- See also: Department Web-site — http://www.uihealthcare.com/depts/med/psychiatry/index.html